CLINICAL TRIAL: NCT05735977
Title: An Open Label Cohort Study Assessing the Near Infrared Fluoroscopic Macro and Microscopic Appearances of Paediatric Renal Parenchyma and Tumours Following Ex-vivo Injection of Indocyanine Green
Brief Title: Nephrogreen. Appearances of Exvivo Renal Tumours Under Near-infrared
Acronym: Nephrogreen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Birmingham Women's and Children's NHS Foundation Trust (Other)
Collaborators: Children's Cancer and Leukaemia Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 22/BC/ONC/NO/655
Record Dates: First submitted 2022-12-20; First posted 2023-02-21 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2024-08

CONDITIONS: Wilms Tumor; Renal Cancer
Keywords: Wilms; Indocyanine Green; Partial Nephrectomy
MeSH Terms: conditions — Wilms Tumor; Kidney Neoplasms

STUDY DESIGN:
Intervention Model Description: Single centre cohort study using consecutive patients. No comparison group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Indocyanine Green (Other): Cohort study using one arm, no comparator group is possible or feasible
  Interventions: Diagnostic Test: Indocyanine Green (ICG)

INTERVENTIONS:
Diagnostic Test: Indocyanine Green (ICG) — Will the use of ICG delineate the margin between normal kidney parenchyma and renal tumour in children at a macroscopic level and can this be replicated at a microscopic level

SUMMARY:
Indocyanine Green (ICG) is a dye which fluoresces under near-infrared (NIR) light. It has been used for several applications in adult surgery. The CI is pioneering its use in children's kidney cancer surgery for lymph node identification and removal. This study concentrates on its use for procedures where only the part of the kidney containing tumour is removed. It is known that kidney tumours in both adults and children do not take up ICG at all. This absence of uptake can be used to define the border between normal and abnormal renal tissue giving a real-time picture of the area of tumour. This then delivers surgeons an intra-operative roadmap for removing only the cancerous part of the kidney. At present the international society of paediatric oncology - renal tumour study group (SIOP-RTSG) protocol, which is followed in the UK, advises consideration of partial nephrectomy for children with bilateral renal tumours and in children with unilateral tumours who have a renal tumour predisposition syndrome. There is ongoing debate about partial nephrectomy in unilateral renal tumour surgery in children who do not have a predisposition syndrome.

This study aims to provide the evidence that paediatric renal tumours do not take up ICG at a naked-eye level and confirm this at a cell level. ICG will be infused into kidneys containing tumour once they have been removed from the patient, The kidney and tumour will be observed under NIR light to show where the areas of fluorescence are. Then, a pathologist will prepare the specimen in theatre, in the same way they would do in the lab. The specimen would be bivalved and reviewed under NIR. Microscopy specimens of the border between normal and abnormal tissue would then be reviewed with an NIR capable microscope. The standard histopathological assessment would then take place.

DETAILED DESCRIPTION:
This study will ascertain if paediatric renal tumours are ICG avid or not. This is critical for determining what the value of using ICG/NIRF will be during nephron sparing surgery (NSS)/ partial nephrectomy in children who have renal tumours that are suitable for this type of surgery. If the normal renal parenchyma is ICG avid but the tumour is not (as has been shown for RCC in adults) then we can conclude that if a fluorescent margin left in-situ on the tumour, then it would be completely resected. Early work at St. Jude has suggested this technique shows promise, but it has not been validated prospectively at a macro or microscopic level.

This is important because in children with unilateral tumours, total nephrectomy has been performed routinely due to concern over leaving behind tumour tissue. If tumour tissue is left behind the patient is upstaged and requires radiotherapy with the consequent sequelae that confers. Radiotherapy to this area invariably damages the kidney so much that it is essentially non-functioning and avoiding this exposure would clearly be ideal. In children with bilateral tumours, retaining as much renal tissue as possible whilst facilitating a complete resection is the goal of surgery. If ICG/NIRF can help with this then it will change the game for this population of patients In addition, this technique will aid in retaining as much normal parenchyma as possible giving the patient better long-term outcomes for renal function. As a further advantage, the study may ascertain if ICG can differentiate between non-cancerous nephrogenic rests (NRs), normal renal parenchyma, and tumour. The difference between these types of tissue is critical when doing NSS because currently only formal histopathological assessment can reliably differentiate NRs from normal tissue or tumour. This is because the definition hinges on whether the lesions have a capsule or not. This is not identifiable on imaging or on core biopsy. The vital feature is that NR's do not require resection, whereas tumour obviously does.

Avidity for ICG may be different in different types of tumours and this will be recorded using the intensity mapping feature of the Storz Rubina Opal1 system. At a cellular level it will be important to investigate why ICG does not cross into tumour and whether this is due to the tumour capsule preventing or limiting vascular flow, or some other factor.

ICG does not affect the histopathological assessment and this research study will validate whether ICG survives the fixing process as this has not been assessed with an NIR capable microscope.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of paediatric renal tumour
* A requirement for radical total nephroureterectomy as part of the treatment

Exclusion Criteria:

* Tumour removed in multiple pieces
* Renal vein thrombus

Ages: 1 Day to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-01-06 (Actual); Study Completion 2025-01-06 (Actual)

PRIMARY OUTCOMES:
Macroscopic appearance | Immediately following tumour resection
  Macroscopic comparison assessment of ICG avidity using Storz Rubina NIR between normal renal parenchyma and tumour.

SECONDARY OUTCOMES:
ICG intensity mapping | Immediately following tumour resection
  Measurement of the quantifiable level of avidity using intensity mapping on a Karl Storz Endoskope™ Opal 1 Rubina system.
Microscopic appearance | Within 2 weeks following tumour resection
  Microscopic comparison of ICG avidity between tumour, non-tumour and nephrogenic rests using a nearinfrared microscope.

CONTACTS AND LOCATIONS:
Overall Officials: Max Pachl, Principal Investigator — Birmingham Women's and Children's NHS Foundation Trust, UK
Locations (1):
- Birmingham children's hospital, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
all IPD that underlie results in a publication

REFERENCES:
- [Background] van den Bos J, Wieringa FP, Bouvy ND, Stassen LPS. Optimizing the image of fluorescence cholangiography using ICG: a systematic review and ex vivo experiments. Surg Endosc. 2018 Dec;32(12):4820-4832. doi: 10.1007/s00464-018-6233-x. Epub 2018 May 18. PMID 29777357
- [Background] Farag S, Frazzini Padilla P, Smith KA, Flyckt R, Sprague ML, Zimberg SE. Fallopian tube perfusion in ex-vivo and in-vivo laparoscopic hysterectomy specimens: potential application for uterine transplantation. Hum Reprod. 2018 Dec 1;33(12):2232-2240. doi: 10.1093/humrep/dey307. PMID 30304437
- [Background] Vujanic GM, Gessler M, Ooms AHAG, Collini P, Coulomb-l'Hermine A, D'Hooghe E, de Krijger RR, Perotti D, Pritchard-Jones K, Vokuhl C, van den Heuvel-Eibrink MM, Graf N; International Society of Paediatric Oncology-Renal Tumour Study Group (SIOP-RTSG). The UMBRELLA SIOP-RTSG 2016 Wilms tumour pathology and molecular biology protocol. Nat Rev Urol. 2018 Nov;15(11):693-701. doi: 10.1038/s41585-018-0100-3. PMID 30310143
- [Background] Dome JS, Fernandez CV, Mullen EA, Kalapurakal JA, Geller JI, Huff V, Gratias EJ, Dix DB, Ehrlich PF, Khanna G, Malogolowkin MH, Anderson JR, Naranjo A, Perlman EJ; COG Renal Tumors Committee. Children's Oncology Group's 2013 blueprint for research: renal tumors. Pediatr Blood Cancer. 2013 Jun;60(6):994-1000. doi: 10.1002/pbc.24419. Epub 2012 Dec 19. PMID 23255438
- [Background] Mitsui Y, Shiina H, Arichi N, Hiraoka T, Inoue S, Sumura M, Honda S, Yasumoto H, Igawa M. Indocyanine green (ICG)-based fluorescence navigation system for discrimination of kidney cancer from normal parenchyma: application during partial nephrectomy. Int Urol Nephrol. 2012 Jun;44(3):753-9. doi: 10.1007/s11255-011-0120-x. Epub 2012 Jan 4. PMID 22215306
- [Background] Soga N, Inoko A, Furusawa J, Ogura Y. Evaluation to Differentiate between Tumor Lesions and the Parenchyma in Partial Nephrectomies for Renal Tumors Based on Quantitative Fluorescence Imaging Using Indocyanine Green Dye. Curr Urol. 2019 Oct;13(2):74-81. doi: 10.1159/000499289. Epub 2019 Oct 1. PMID 31768173
- [Background] Mrad C, Coulomb-Lhermine A, Tabone MD, Ulinski T, Audry G, Irtan S. Evaluation of the nephron-sparing surgery formula in Wilms tumors. Pediatr Blood Cancer. 2020 Dec;67(12):e28661. doi: 10.1002/pbc.28661. Epub 2020 Aug 18. PMID 32808461
- [Background] Rickard M, Fernandez N, Blais AS, Shalabi A, Amirabadi A, Traubici J, Lee W, Gleason J, Brzezinski J, Lorenzo AJ. Volumetric assessment of unaffected parenchyma and Wilms' tumours: analysis of response to chemotherapy and surgery using a semi-automated segmentation algorithm in children with renal neoplasms. BJU Int. 2020 May;125(5):695-701. doi: 10.1111/bju.15026. Epub 2020 Feb 27. PMID 32012416
- [Background] Cozzi DA, Ceccanti S, Frediani S, Schiavetti A, Cozzi F. Chronic kidney disease in children with unilateral renal tumor. J Urol. 2012 May;187(5):1800-5. doi: 10.1016/j.juro.2011.12.109. Epub 2012 Mar 17. PMID 22424685
- [Background] Cozzi DA, Ceccanti S, Cozzi F. Renal function up to the 5th decade of life after nephrectomy in childhood: A literature review. Nephrology (Carlton). 2018 May;23(5):397-404. doi: 10.1111/nep.13202. PMID 29194872
- [Background] Green DM, Wang M, Krasin MJ, Davidoff AM, Srivastava D, Jay DW, Ness KK, Shulkin BL, Spunt SL, Jones DP, Lanctot JQ, Shelton KC, Brennan RC, Mulrooney DA, Ehrhardt MJ, Gibson TM, Kurt BA, Robison LL, Hudson MM. Long-term renal function after treatment for unilateral, nonsyndromic Wilms tumor. A report from the St. Jude Lifetime Cohort Study. Pediatr Blood Cancer. 2020 Oct;67(10):e28271. doi: 10.1002/pbc.28271. Epub 2020 Jul 24. PMID 32706494
- [Background] Tan XH, Zhang DY, Liu X, Lin T, He DW, Li XL, Wei GH. Retrospective analysis to determine outcomes of patients with bilateral Wilms tumor undergoing nephron sparing surgery: 15-year tertiary single-institution experience. Pediatr Surg Int. 2018 Apr;34(4):427-433. doi: 10.1007/s00383-018-4232-6. Epub 2018 Jan 24. PMID 29368077
- [Background] Kieran K, Williams MA, Dome JS, McGregor LM, Krasin MJ, Davidoff AM. Margin status and tumor recurrence after nephron-sparing surgery for bilateral Wilms tumor. J Pediatr Surg. 2013 Jul;48(7):1481-5. doi: 10.1016/j.jpedsurg.2013.02.033. PMID 23895958